CLINICAL TRIAL: NCT06101537
Title: Correlation Patterns of Brain Temperature-Pressure in Acute Brain Injury：a Multicenter Prospective Cohort Study, MERCURY
Brief Title: Correlation Patterns of Brain Temperature-Pressure in Acute Brain Injury
Acronym: MERCURY
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HX-B-2023067
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intracranial Pressure; Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Hemorrhage
Keywords: brain temperature monitoring; intracranial pressure monitoring; severe brain injury; subarachnoid hemorrhage; cerebral hemorrhage; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Hemorrhage; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brain temperature-pressure monitoring group: From a neurointensive care unit with intracranial pressure monitoring during treatment, which allows continuous recording of brain temperature-pressure data, in patients with moderate and severe acute brain injury due to subarachnoid hemorrhage, cerebral hemorrhage, and craniocerebral trauma.
  Interventions: Device: Brain temperature-pressure monitoring

INTERVENTIONS:
Device: Brain temperature-pressure monitoring — An intracranial pressure monitoring device that continuously records brain temperature-pressure data was used during treatment.

SUMMARY:
The goal of this prospective, multicenter, observational, cohort trail is to explore the pattern of brain temperature-brain pressure association in acute brain injury and to clarify its predictive value for prognosis and neurological function 30 days after acute brain injury.

DETAILED DESCRIPTION:
Temperature abnormalities have long been recognized as signs of disease. Brain temperature, as part of body temperature, reflects body temperature and brain metabolism during physiologic states. There is growing evidence that brain cell function is unequivocally temperature dependent and that brain temperature after brain injury cannot be reliably predicted by core body temperature. Brain temperature is therefore increasingly becoming an important alternative to brain pressure, enabling patients with a variety of brain injuries to benefit from continuous brain temperature monitoring. Meanwhile, the correlation between intracranial pressure, which is currently the most widely used indicator in clinical practice, and brain temperature in patients with acute brain injury remains unelucidated. Whether the correlation between brain temperature and intracranial pressure has certain patterns and rhythms that can indirectly reflect the brain function of patients under the condition of injury and have a predictive value for clinical outcomes is the main research objective of this study. It is hoped that the present study will explore the correlation between brain temperature and brain pressure and the pattern of the correlation, as well as its impact on clinical prognosis. It provides a more precise target for intervention to further improve the prognosis of patients with acute brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, male or female, 18 to 65 years of age;
2. Acute brain injury due to subarachnoid hemorrhage, cerebral hemorrhage, or craniocerebral trauma;
3. Glasgow Coma Scale (GCS) score of 3-12;
4. Have undergone intracranial pressure monitoring probe placement, which allows continuous recording of brain temperature and pressure data;
5. Signed informed consent.

Exclusion Criteria:

1. GCS ≥13 points;
2. Patients with concomitant intracranial infections, cerebral ischemia, congenital malformations, autoimmune encephalitis, or craniocerebral tumors;
3. At the time of onset, there was a combination of systemic malignant tumor, acute stage of major systemic organ disease, or stage of functional decompensation;
4. Maternity;
5. Undergoing experimental drug or instrumental trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe acute brain injury due to subarachnoid hemorrhage, cerebral hemorrhage, and craniocerebral trauma from 20 centers with intracranial pressure monitoring during treatment, which allows continuous recording of brain temperature-brain pressure data.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Correlation Patterns of brain temperature-brain pressure in acute brain injury | At baseline and on days 1-7 after receiving brain temperature-brain pressure monitoring
  By using a brain temperature-pressure monitoring device, the correlation was analyzed by continuously recording brain temperature-pressure data and plotting time-brain temperature and time-brain pressure curves in patients with moderate and severe acute brain injury due to subarachnoid hemorrhage, cerebral hemorrhage, and craniocerebral trauma.
Predictive value of brain temperature-brain pressure correlation patterns on prognosis and neurological function in patients with acute brain injury | 30 days after acute brain injury
  Predictive value of the brain temperature-brain pressure correlation patterns on the prognosis and neurological function of patients after acute brain injury as clarified by patients' Extended Glasgow Outcome Scale (GOSE) (an 8-point scale, ranging from death to "upper good recovery" ).

SECONDARY OUTCOMES:
Rhythmic patterns of brain temperature in acute brain injury | At baseline and on days 1-7 after receiving brain temperature-brain pressure monitoring
  To explore the rhythmic pattern of brain temperature in acute brain injury by using a brain temperature-pressure monitoring device, obtaining continuous brain temperature data, and plotting the brain temperature-time curve.
Predictive value of brain temperature rhythmic patterns on prognosis and neurological function in patients with acute brain injury | 30 days after acute brain injury
  Predictive value of the brain temperature rhythmic patterns on the prognosis and neurological function of patients after acute brain injury as clarified by patients' Extended Glasgow Outcome Scale (GOSE) (an 8-point scale, ranging from death to "upper good recovery" )
Differences in brain temperature-brain pressure correlation patterns by injury type | At baseline and on days 1-7 after receiving brain temperature-brain pressure monitoring
  By using a brain temperature-brain pressure monitoring device, brain temperature-brain pressure data were continuously recorded in patients with moderate and severe acute brain injuries due to subarachnoid hemorrhage, cerebral hemorrhage, and craniocerebral trauma. And time-brain temperature and time-brain pressure curves were plotted to analyze the differences between different injury types.
Number of participants with brain temperature-pressure-related adverse events | At baseline and on days 1-7 after receiving brain temperature-brain pressure monitoring
  After obtaining the predictive value of the brain temperature-pressure correlation patterns for prognosis and neurological function in patients with acute brain injury, the number of participants with associated adverse events was assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Guoyi Gao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weng WJ, Yang C, Huang XJ, Zhang YM, Liu JF, Yao JM, Zhang ZH, Wu XS, Mei T, Zhang CD, Jia J, Shi XF, Mao Q, Feng JF, Gao GY, Jiang JY. Effects of Brain Temperature on the Outcome of Patients with Traumatic Brain Injury: A Prospective Observational Study. J Neurotrauma. 2019 Apr 1;36(7):1168-1174. doi: 10.1089/neu.2018.5881. Epub 2018 Oct 10. PMID 30215286